CLINICAL TRIAL: NCT05380882
Title: A Phase I Study of TQB2930 Injection in Patients With Advanced Cancers
Brief Title: Clinical Trial of the TQB2930 Injection in Patients With Advanced Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2930-I-01
Record Dates: First submitted 2022-05-06; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Advanced Cancers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2930 injection (Experimental): Drug:Weekly intravenous infusion of TQB2930 injection,21 days as a treatment cycle. (2.5mg/kg, 5mg/kg, 10mg/kg) Drug:Every two weeks intravenous infusion of TQB2930 injection , 28 days as a treatment cycle.(20mg/kg) Drug:Every three weeks intravenous infusion of TQB2930 injection, 21 days as a treatment cycle. (30mg/kg)
  Interventions: Drug: TQB2930 injection

INTERVENTIONS:
Drug: TQB2930 injection — TQB2930 is an anti-HER2 bispecific antibody.

SUMMARY:
TQB2930 is an anti-HER2 (Human Epidermal Growth Factor Receptor 2) bispecific antibody that can simultaneously bind two epitopes of HER2, leading to a dual HER2 signal blockage. This is a phase I study to evaluate the safety, tolerability and effectiveness of TQB2930 injection in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1 Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* 2 Male or female patient 18 to 75 years of age, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and life expectancy ≥12 weeks;
* 3 Histologically or cytologically confirmed, locally advanced tumors, Priority will be given to subjects with HER2 positive solid tumor;
* 4 Malignant tumor that failed from standard treatment or had no standard treatment;
* 5 According to the RECIST 1.1 standard, patient with at least one evaluable lesion;
* 6 The main organs function well;
* 7 Male or female patient had no plans to become pregnant and voluntarily took effective contraceptive measures from agree with the study to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* 1 Concurrent secondary malignancy. or other malignancy with no evidence of disease for more than 3 years;
* 2 History of uncontrolled intercurrent illness;
* 3 Major surgical procedure, radiotherapy, chemotherapy, or immunotherapy within 4 weeks prior to first dose;
* 4 Patients with known symptomatic brain metastases;
* 5 Receiving any other investigational agent within 4 weeks before first dose;
* 6 Unstable or serious concurrent medical conditions, as assessed by the Investigators, that would substantially increase the risk-benefit ratio of participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 or 28 days)
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI CTCAE v5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred from the first dose to the end of the first treatment cycle.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 21 or 28 days).
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Adverse events (AE) rate | From date of the first dose until the date of 28 days after last dose or new anti-tumor treatment, whichever came first.
  The occurrence and severity of all AEs

SECONDARY OUTCOMES:
immunogenicity | Cycle 1 Day 1, Cycle 2 Day1, Cycle 4 Day1, Cycle 7 Day1, Cycle 12 Day1: pre-dose and end of the infusion.(each cycle is 21 or 28 days)
  Incidence of anti-drug antibody (ADA)
Pharmacokinetics: The area under the curve (AUC) | Cycle1Day1, Cycle1Day8, Cycle1Day815, Cycle2 Day1, Cycle2Day8, Cycle2Day15 and Cycle3Day1: pre-dose, Cycle1Day1:at 0.5, 4, 8, 24, 48, 72, and 240 hours after infusion. Cycle2Day1:at 0.5, 4, 8, 24, 48, 72, and 240 hours after infusion.(21 or 28 days each)
  The area under the curve (AUC) of serum concentration of TQB2930
Pharmacokinetics:Peak concentration (Cmax) | Cycle1Day1, Cycle1Day8, Cycle1Day815, Cycle2 Day1, Cycle2Day8, Cycle2Day15 and Cycle3Day1: pre-dose, Cycle1Day1:at 0.5, 4, 8, 24, 48, 72, and 240 hours after infusion. Cycle2Day1:at 0.5, 4, 8, 24, 48, 72, and 240 hours after infusion.21 or 28 days each
  Maximum observed concentration (Cmax) of TQB2930
Pharmacokinetics: T1/2 | Cycle1Day1, Cycle1Day8, Cycle1Day815, Cycle2 Day1, Cycle2Day8, Cycle2Day15 and Cycle3Day1: pre-dose, Cycle1Day1:at 0.5, 4, 8, 24, 48, 72, and 240 hours after infusion. Cycle2Day1:at 0.5, 4, 8, 24, 48, 72, and 240 hours after infusion.21 or 28 days each
  Terminal half-life (T1/2)
Objective Response Rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100weeks
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria
Disease control rate (DCR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100weeks
  Defined as the proportion of subjects with CR, PR, or SD (Stable Disease).
Duration of Response (DOR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100weeks
  Defined as the time from first documented response to documented disease progression.
Progression-free survival (PFS) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100weeks
  Defined as the time from the first dose of TQB2928 to the first occurrence of disease progression or death from any cause.
Overall survival(OS) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100weeks
  Overall survival refers to the time from the first treatment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China